CLINICAL TRIAL: NCT06824181
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, 4-arm Study to Investigate the Mixed Vaccination Schedules of a 21-valent Pneumococcal Conjugate Vaccine and a 20-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers
Brief Title: Study of Mixed Vaccination Schedules With a 21-valent Pneumococcal Conjugate Vaccine and a 20-valent Pneumococcal Conjugate Vaccine in Healthy Infants From Approximately 2 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK00031; U1111-1294-7911 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Immunization
MeSH Terms: interventions — RIX4414 vaccine; RotaTeq; Vaxelis; Chickenpox Vaccine; Measles-Mumps-Rubella Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind
  * Blinding for vaccine group assignment: participants and participant's parent(s) / legally acceptable representative(s) (LARs), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: those preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 20vPCV-PCV21-PCV21-PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 4-dose 20vPCV regimen at approximately 2 MoA, PCV21 at 4 MoA, PCV21 at 6 MoA and PCV21 at 12 to 15 MoA
  Interventions: Biological: PCV21 vaccine; Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix
- Group 2: 20vPCV-20vPCV-PCV21-PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 4-dose 20vPCV regimen at approximately 2 MoA, 20vPCV at 4 MoA, PCV21 at 6 MoA and PCV21 at 12 to 15 MoA
  Interventions: Biological: PCV21 vaccine; Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix
- 20vPCV-20vPCV-20vPCV-PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 4-dose 20vPCV regimen at approximately 2 MoA, 20vPCV at 4 MoA, 20vPCV at 6 MoA and PCV21 at 12 to 15 MoA
  Interventions: Biological: PCV21 vaccine; Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix
- 20vPCV-20vPCV-20vPCV-20vPCV (Active Comparator): Participants will be administered via intramuscular injection (IM) a 4-dose 20vPCV regimen at approximately 2 MoA, 20vPCV at 4 MoA, 20vPCV at 6 MoA and 20vPCV at 12 to 15 MoA
  Interventions: Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: Rotarix; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Priorix; Biological: VAQTA; Biological: Havrix

INTERVENTIONS:
Biological: PCV21 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: 515
  Arms: 20vPCV-20vPCV-20vPCV-PCV21; Group 1: 20vPCV-PCV21-PCV21-PCV21; Group 2: 20vPCV-20vPCV-PCV21-PCV21
Biological: Prevnar 20 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Prevnar20™
Biological: M-M-R II vaccine — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: M-M-R™ II
Biological: Rotarix — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: Rotarix™
Biological: RotaTeq — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: RotaTeq™
Biological: Vaxelis vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Vaxelis™
Biological: Varivax — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: Varivax™
Biological: Priorix — Pharmaceutical form:Lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous
  Other Names: Priorix™
Biological: VAQTA — Pharmaceutical form:Suspension for Injection-Route of administration:Intramuscular
  Other Names: VAQTA™
Biological: Havrix — Pharmaceutical form:Suspension for Injection-Route of administration:Intramuscular
  Other Names: Havrix™

SUMMARY:
This study is a Phase 3, randomized, modified double-blind study which aims to measure whether the investigational pneumococcal conjugate vaccine PCV21 is safe and can help the body to develop germ-fighting agents called "antibodies" (immunogenicity) when it is given after 1 dose, 2 doses, or 3 doses of a licensed 20-valent pneumococcal vaccine compared to when 20-valent pneumococcal vaccine is given as a complete series in infants aged from approximately 2 months (42 to 89 days).

The study duration per participant will be up to approximately 19 months. The study vaccines (either PCV21 or 20vPCV) will be administered at approximately 2, 4, 6 and 12 to 15 months of age (MoA). Routine pediatric vaccines will be given as per local recommendations.

There will be 6 study visits:

Visit (V)01, V02 separated from V01 by 60 days, V03 separated from V02 by 60 days, V04 separated from V03 by 30 days, V05 at 12 months of age until 15 months of age, V06 separated from V05 by 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 89 days on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable as assessed by the investigator

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed Streptococcus pneumoniae infection or disease.
* History of seizure or significant stable or progressive neurologic disorders such as inflammatory nervous system diseases, encephalopathy, cerebral palsy
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Thrombocytopenia, or known thrombocytopenia, as reported by the parent/legal acceptable representative (LAR), contraindicating intramuscular (IM) injection.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Previous vaccination against Streptococcus pneumoniae
* Receipt of immune globulins, blood or blood-derived products since birth
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 580 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Presence of any immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Number of participants experiencing solicited and unsolicited immediate AEs
Presence of solicited injection site and systemic reactions through 7 days after each vaccine injection | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site and systemic reactions
Presence of unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs through 30 days after each vaccine injection | Through 30 days after each vaccine injection
  Number of participants experiencing unsolicited injection site reactions and unsolicited systemic AEs
Presence of serious adverse events (SAEs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 19 months
  Number of participants experiencing SAEs
Presence adverse events of special interest (AESIs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 19 months
  Number of participants experiencing AESIs
Serotype Specific IgG GMCs for Each Pneumococcal Serotype at 30 Days PD4 | 30 days PD4
  The GMCs for serotype-specific pneumococcal IgG antibodies are measured using electro-chemiluminescence assay (ECL)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (17):
  - Kaiser Permanente Los Angeles Medical Center- Site Number : 8400025, Los Angeles, California
  - The Medici Medical Research- Site Number : 8400008, Hollywood, Florida
  - Clinsearch Inc at Dr. Gala, LLC- Site Number : 8400027, Miami, Florida
  - Atlantis Clinical Research, LLC- Site Number : 8400009, Miami, Florida
  - Velocity Clinical Research, Sioux City- Site Number : 8400007, Sioux City, Iowa
  - Michael W. Simon, M.D., PSC- Site Number : 8400001, Lexington, Kentucky
  - Velocity Clinical Research New Orleans- Site Number : 8400006, New Orleans, Louisiana
  - Finger Lakes Medical Research, PLLC- Site Number : 8400022, Cortland, New York
  - University of Rochester Medical Center- Site Number : 8400019, Rochester, New York
  - ~SUNY Upstate Medical University- Site Number : 8400015, Syracuse, New York
  - Kid's Way Pediatrics- Site Number : 8400013, Hermitage, Pennsylvania
  - Carolina Family Care- Site Number : 8400014, Charleston, South Carolina
  - Helios- Site Number : 8400016, Burleson, Texas
  - Clinsearch Inc at VAST Clinical Research- Site Number : 8400028, Euless, Texas
  - Kool Kids Pediatrics- Site Number : 8400012, Houston, Texas
  - University of Texas Medical Branch- Site Number : 8400005, League City, Texas
  - Javara Inc/Privia Medical Group North Texas, PLLC- Site Number : 8400024, Stephenville, Texas
- Chile (3):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago
- Mexico (4):
  - Investigational Site Number : 4840003, León, Guanajuato
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840002, Temixco, Morelos
  - Investigational Site Number : 4840004, Tlaltizapán, Morelos
- Philippines (3):
  - Investigational Site Number : 6080001, Cebu
  - Investigational Site Number : 6080002, Quezon
  - Investigational Site Number : 6080003, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PSK00031 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26406&tenant=MT_SNY_9011